CLINICAL TRIAL: NCT00013000
Title: A Multi-Site Study of Strategies for Implementing Schizophrenia Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPG 97-027
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Test strategy for implementation guideline

INTERVENTIONS:
Behavioral: Test strategy for implementation guideline

SUMMARY:
Schizophrenia, a chronic psychiatric disorder, is the second most frequent VA discharge diagnosis. Medication management practices for schizophrenia often are not guideline-concordant and place patients at risk for adverse outcomes. This project tests a new strategy to standard implementation for VHA Schizophrenia Guidelines.

DETAILED DESCRIPTION:
Background:

Schizophrenia, a chronic psychiatric disorder, is the second most frequent VA discharge diagnosis. Medication management practices for schizophrenia often are not guideline-concordant and place patients at risk for adverse outcomes. This project tests a new strategy to standard implementation for VHA Schizophrenia Guidelines.

Objectives:

Research objectives are: (1) to compare the effectiveness of a conceptually-based, enhanced intervention to that of a basic educational strategy with regard to improving guideline adherence and patient compliance; (2) to compare the effectiveness of the two strategies with regard to improving symptom and side effect outcomes; (3) to determine the effect of the enhanced intervention on service utilization for acute exacerbations of schizophrenia; (4) to determine the extent to which guideline-concordant medication management improves patient outcomes; and (5) to examine providers' knowledge of and attitudes toward guidelines.

Methods:

Thirteen VA sites were considered for the study, and VistA data were extracted to assess baseline guideline performance. Seven sites were selected and received basic education about schizophrenia guidelines. Three of these sites were randomly selected to receive the enhanced intervention, employing a nurse coordinator to promote providers' guideline adherence and patients' treatment adherence. Subjects with an acute exacerbation of schizophrenia were enrolled and were interviewed at baseline and six months using the Positive and Negative Syndrome Scale, the Schizophrenia Outcomes Module, and the Barnes Akathisia Scale. Data on guideline adherence were collected from medical records and VistA files. When data collection is completed, analyses will be conducted to determine the effectiveness of the enhanced intervention with regard to improving guideline adherence and patient outcomes.

Status:

The project is ongoing. To date, 401 subjects have been enrolled in the intervention study. The rate of completed follow-up assessments to date is 86 percent.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a diagnosis of schizophrenia. 2. Subjects must have been admitted to an inpatient psychiatry unit or seen in an ambulatory care clinic or the Emergency Room at a study site for symptoms of acute exacerbation. 3. Must be able to provide informed consent themselves or informed consent by a guardian.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Owen, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (6):
- United States (6):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Maryland
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

REFERENCES:
- [Result] Hamilton J, Guthrie E, Creed F, Thompson D, Tomenson B, Bennett R, Moriarty K, Stephens W, Liston R. A randomized controlled trial of psychotherapy in patients with chronic functional dyspepsia. Gastroenterology. 2000 Sep;119(3):661-9. doi: 10.1053/gast.2000.16493. PMID 10982759
- [Result] Owen RR, Hudson T, Thrush C, Thapa P, Armitage T, Landes RD. The effectiveness of guideline implementation strategies on improving antipsychotic medication management for schizophrenia. Med Care. 2008 Jul;46(7):686-91. doi: 10.1097/MLR.0b013e3181653d43. PMID 18580387